CLINICAL TRIAL: NCT00119756
Title: A Randomized, Crossover Study to Evaluate the Overall Safety and Tolerability of Paliperidone Palmitate Injected in the Deltoid or Gluteus Muscle in Patients With Schizophrenia
Brief Title: A Safety and Tolerability Study of Paliperidone Palmitate Injected in the Shoulder or the Buttock Muscle in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR002350
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Intramuscular injection; Deltoid muscle; Gluteus muscle; Paliperidone palmitate
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone palmitate

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of intramuscular injections (to the buttocks or to the shoulders) of paliperidone palmitate in patients with schizophrenia.

DETAILED DESCRIPTION:
To date, all prior trials involving intramuscular injection of paliperidone palmitate were conducted with buttock administration. This is a randomized, multicenter, crossover design study in evaluating safety and tolerability of paliperidone palmitate in two different injection sites. The study hypothesis is that there will be no difference in safety and tolerability between buttock injection compared to shoulder injection at any of the three different doses of paliperidone palmitate. The patients will receive intramuscular injections of paliperidone palmitate in either their buttocks or in their shoulders

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed an informed consent
* The patient must meet the diagnostic criteria for schizophrenia
* Female patient must be postmenopausal for at least 2 years or have negative pregnancy test result at screening
* The patient must be able to perform study requirements (e.g. answer questionnaire)

Exclusion Criteria:

* Primary, active diagnosis other than schizophrenia
* Psychiatric inpatient hospitalization for relapse of symptoms of schizophrenia in the past 90 days
* Change in their antipsychotic medication in the past 45 days
* Diagnosis of active substance dependence within 3 months
* History of treatment resistance
* History of concurrent significant or unstable diseases (e.g. heart, lung, or liver diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2005-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Safety evaluation (e.g. incidence of adverse events) between start and finish of the trial

SECONDARY OUTCOMES:
Pharmacokinetic evaluations (e.g. blood level of the drug) at finish of trial; Efficacy measures at finish of trial

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Hough D, Lindenmayer JP, Gopal S, Melkote R, Lim P, Herben V, Yuen E, Eerdekens M. Safety and tolerability of deltoid and gluteal injections of paliperidone palmitate in schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Aug 31;33(6):1022-31. doi: 10.1016/j.pnpbp.2009.05.014. Epub 2009 May 28. PMID 19481579
- See also: A safety and tolerability study of paliperidone palmitate injected in the deltoid or the gluteal muscle in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=469&filename=CR002350_CSR.pdf